# CHARACTERISTICS OF MENSTRUAL CYCLE IN HEALTHCARE PROFESSIONALS AT COVID 19 PANDEMIC HOSPITAL

HNEAH KAEK 2020/KK/10

Sevcan Arzu ARINKAN-2020-05-03T22\_54\_16

May 2020

STUDY PROTOCOL

### **OBJECTIVES**

The COVID-19 pandemic has impacted healthcare workers physically and psychologically. Healthcare workers have ben required to work under stressful conditions and take difficult decisions involving ethical implications. Increasing work demands on healthcare professionals conflict with their duties to family and friends, which causes psychological stress. All of these factors may negatively affect their menstrual cycle.

The aim of this study is to examine whether there is a change in menstrual cycle characteristics during pandemia. Also, we aim to investigate whether there is an association between covid infection and menstrual cycle changes.

### **DESIGN**

Healthy females who are working at Covid 19 clinic at least 1 month, are included to study. After informed consent, detailed information are collected using structured questionnaires about their reproductive factors and menstrual cycles.

### **METHODS**

This cross-sectional study is conducted with healthy female participants who are working at Covid 19 pandemic clinics at Haydarpasa Numune Research and Training Hospital in Turkey. Only participants who are sure about their pertinant information are enrolled in the study. Detailed information is collected using structured questionnaires by face to face.

Primary Outcome Measure:

- 1. Irregular menstrual cycle
- 1 month after starting to work at pandemic clinic
- 2.Length of cycle (day)
- 1 month after starting to work at pandemic clinic
- 3. Duration of bleeding (day)
- 1 month after starting to work at pandemic clinic
- 4. Amount of flow (number of used tampons)
- 1 month after starting to work at pandemic clinic
- 5. Dysmenorrhea status (VAS score)
- 1 month after starting to work at pandemic clinic

## Secondary Outcome Measures:

1. Length of cycle difference between covid positive and negative healthcare workers

First menstrual period after covid infection

2.Duration of bleeding difference between covid positive and negative healthcare workers First menstrual period after covid infection]

3.Amount of flow difference between covid positive and negative healthcare workers First menstrual period after covid infection

Inclusion Criteria:

Working at Covid 19 Pandemic Hospital
Being at between 18 and 47 years old
Having menstruation

**Exclusion Criteria:** 

Oral contraceptive users

**Pregnants** 

Having malignancy

Having primary amenorrhea

Being at menopause

Lactation

Statistical Analysis Plan

The study was approved by the Ethics and Clinical Investigation Committee. Statistical Package for the Social Sciences (SPSS; Version 20.0, Chicago, IL, USA) will be used for statistical analyses. Descriptive statistics will be presented as mean ± standard deviation (SD) for normally distributed data, and as counts and percentages for categorical data. The relationship between the categorical variables will be examined using the Chi-square test and Fisher Exact Test. Results will be evaluated with a confidence interval of 95%, and p<0.05/p<0,01 will be considered statistically significant. Kolmogorov-Smirnov test will be used for the assessment of the normality of data. Mann- Whitney U test will be used for the data not normally distributed.